CLINICAL TRIAL: NCT07267130
Title: Phase I Clinical Study to Evaluate the Safety, Tolerability and Pharmacokinetic Profile of TQC3302 Inhalation Spray in Healthy Adult Subjects in China
Brief Title: A Clinical Study to Evaluate the Safety, Tolerability and Pharmacokinetic Profile of TQC3302 Inhalation Spray in Healthy Adult Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical (Guangzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TQC3302-I-01
Record Dates: First submitted 2025-11-25; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Inhalation; Tiotropium Bromide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- TQC3302 inhalation spray (50/2.5/2.5μg) (Experimental): Administered as a single dose
  Interventions: Drug: TQC3302 inhalation spray
- TQC3302/Spiolto® Respimat® /Pulmicort® (Experimental): Each drug is administered as a single dose.
  TQC3302 inhalation spray (50/2.5/2.5μg); TQC3302 inhalation spray (100/2.5/2.5μg); Spiolto® Respimat® : Tiotropium bromide and olodaterol hydrochloride inhalation spray (2.5/2.5μg); Pulmicort® : Budesonide Powder for Inhalation (200μg)
  Interventions: Drug: TQC3302 inhalation spray+ TQC3302 inhalation spray+Tiotropium bromide and olodaterol hydrochloride inhalation spray +Budesonide Powder for Inhalation
- TQC3302/Pulmicort®/Spiolto® Respimat® (Experimental): Each drug is administered as a single dose.
  TQC3302 inhalation spray (100/2.5/2.5μg); Spiolto® Respimat®: Tiotropium bromide and olodaterol hydrochloride inhalation spray (2.5/2.5μg) ; Pulmicort®: Budesonide Powder for Inhalation (200μg) TQC3302 inhalation spray (50/2.5/2.5μg)
  Interventions: Drug: TQC3302 inhalation spray+Tiotropium bromide and olodaterol hydrochloride inhalation spray +Budesonide Powder for Inhalation+ TQC3302 inhalation spray
- TQC3302/Spiolto® Respimat®/Pulmicort® (Experimental): Each drug is administered as a single dose.
  Spiolto® Respimat®: Tiotropium bromide and olodaterol hydrochloride inhalation spray (2.5/2.5μg); Pulmicort® : Budesonide Powder for Inhalation (200μg); TQC3302 inhalation spray (50/2.5/2.5μg); TQC3302 inhalation spray (100/2.5/2.5μg)
  Interventions: Drug: Tiotropium bromide and olodaterol hydrochloride inhalation spray +Budesonide Powder for Inhalation+ TQC3302 inhalation spray+ TQC3302 inhalation spray
- Spiolto® Respimat® /Pulmicort®/TQC3302 (Experimental): Each drug is administered as a single dose.
  Pulmicort®: Budesonide Powder for Inhalation (200μg); TQC3302 inhalation spray (50/2.5/2.5μg); TQC3302 inhalation spray (100/2.5/2.5μg); Spiolto® Respimat®: Tiotropium bromide and olodaterol hydrochloride inhalation spray (2.5/2.5μg)
  Interventions: Drug: Budesonide Powder for Inhalation+ TQC3302 inhalation spray+ TQC3302 inhalation spray+ Tiotropium bromide and olodaterol hydrochloride inhalation spray
- TQC3302 inhalation spray (200/5/5μg)-single dose (Experimental): TQC3302 inhalation spray is administered as a single dose.
  Interventions: Drug: TQC3302 inhalation spray
- TQC3302 inhalation spray (100/5/5μg) (Experimental): Single dose during Day 1-Day 7
  Interventions: Drug: TQC3302 inhalation spray
- TQC3302 inhalation spray (200/5/5μg) (Experimental): Single dose during Day 1-Day 7
  Interventions: Drug: TQC3302 inhalation spray

INTERVENTIONS:
Drug: TQC3302 inhalation spray — TQC3302 inhalation spray is a targeted inhibitor
  Arms: TQC3302 inhalation spray (100/5/5μg); TQC3302 inhalation spray (200/5/5μg); TQC3302 inhalation spray (200/5/5μg)-single dose; TQC3302 inhalation spray (50/2.5/2.5μg)
Drug: TQC3302 inhalation spray+ TQC3302 inhalation spray+Tiotropium bromide and olodaterol hydrochloride inhalation spray +Budesonide Powder for Inhalation — TQC3302 inhalation spray is a targeted inhibitor, Tiotropium bromide and olodaterol hydrochloride inhalation spray is a targeted inhibitor, Budesonide Powder for Inhalation is a Inhaled Corticosteroids.
  Arms: TQC3302/Spiolto® Respimat® /Pulmicort®
Drug: TQC3302 inhalation spray+Tiotropium bromide and olodaterol hydrochloride inhalation spray +Budesonide Powder for Inhalation+ TQC3302 inhalation spray — TQC3302 inhalation spray is a targeted inhibitor, Tiotropium bromide and olodaterol hydrochloride inhalation spray is a targeted inhibitor, Budesonide Powder for Inhalation is a Inhaled Corticosteroids.
  Arms: TQC3302/Pulmicort®/Spiolto® Respimat®
Drug: Tiotropium bromide and olodaterol hydrochloride inhalation spray +Budesonide Powder for Inhalation+ TQC3302 inhalation spray+ TQC3302 inhalation spray — TQC3302 inhalation spray is a targeted inhibitor, Tiotropium bromide and olodaterol hydrochloride inhalation spray is a targeted inhibitor, Budesonide Powder for Inhalation is a Inhaled Corticosteroids.
  Arms: TQC3302/Spiolto® Respimat®/Pulmicort®
Drug: Budesonide Powder for Inhalation+ TQC3302 inhalation spray+ TQC3302 inhalation spray+ Tiotropium bromide and olodaterol hydrochloride inhalation spray — TQC3302 inhalation spray is a targeted inhibitor, Tiotropium bromide and olodaterol hydrochloride inhalation spray is a targeted inhibitor, Budesonide Powder for Inhalation is a Inhaled Corticosteroids.
  Arms: Spiolto® Respimat® /Pulmicort®/TQC3302

SUMMARY:
Healthy adult subjects were selected to use TQC3302 inhalation spray to evaluate the safety, tolerability, and pharmacokinetic characteristics of single and multiple inhalations of TQC3302 inhalation spray in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Subjects voluntarily joined the study, sign informed consent form before the study and fully understand the study content
* Healthy subjects aged between 18 and 55 years (inclusive),both male and female
* The male subject should weigh at least 50kg, the female subject should weigh at least 45kg. And body mass index (BMI) within 19~28 kg/m2
* Inhalation administration training qualified.
* During the screening period, the percentage of predicted value for forced expiratory volume in one second (FEV1) before bronchodilator administration is ≥80%, and FEV1/forced vital capacity (FVC) is ≥70%.
* Have no pregnancy plan and voluntarily take effective contraception measures from time of screening to at least 90 days after the last dose (subjects and their partners)

Exclusion Criteria:

* Individuals with a history of glaucoma, functional constipation, benign prostatic hyperplasia, urinary tract obstruction, etc
* Current history of active tuberculosis, bronchiectasis or other non-specific lung diseases
* People who have received or are planning to receive inactive or active vaccines during the 30 days prior to the screening period and the entire study period
* Any history of drug allergies, Individuals with a specific history of allergies or allergies
* Had undergone surgery within 1 month prior to screening period or expected to undergo surgery during the study period
* People with special dietary requirements who cannot follow a standard diet;
* People who have potential difficulty in blood collection, or have a history of halo needles or blood sickness；
* History of drug or narcotics abuse or a positive result of urine drug test at screening
* People who have abnormal and clinically significant results in vital signs, physical examination, laboratory tests, Chest radiograph and abdominal ultrasound during screening period
* Subjects Positive for Any of Hepatitis B Virus Surface Antigen (HBsAg), Hepatitis C Virus Antibody (Anti-HCV), Human Immunodeficiency Virus Antibody (Anti-HIV), and Treponema Pallidum Antibody (Anti-TP)
* Pregnant or lactating women or those with positive blood pregnancy test results during the screening period

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Treatment Emergent Adverse Event | From the use of the investigational drug until the last study visit, up to Day 14
  The incidence and severity of adverse events after treatment From the use of the investigational drug until the last study visit.
The subject with abnormal security check | From the use of the investigational drug until the last study visit, up to Day 14
  The frequency, incidence, and severity of laboratory tests, vital signs, physical examinations, electrocardiogram examinations, etc.

SECONDARY OUTCOMES:
Cmax after dose | Single dose：pre-dose, at 2,5,8,12,25,45 minutes,1,2,4,8,12,24, 48,72,120 hours after-dose (When using Budesonide Powder for Inhalation, there is no need to monitor at 48, 72, and 120 hours after the end of administration)
  The Cmax is the maximum observed plasma concentration of study drug
Area Under the Concentration-Time Curve From 0 to Last Observation (AUC [0-t]) | Single dose：pre-dose, at 2,5,8,12,25,45 minutes,1,2,4,8,12,24, 48,72,120 hours after-dose (When using Budesonide Powder for Inhalation, there is no need to monitor at 48, 72, and 120 hours after the end of administration)
  To characterize the pharmacokinetics of TQC3302 by assessment of area under the plasma concentration time curve from the first dose to a certain time point
Area Under the Concentration-Time Curve From Zero to Infinity (AUC [0-infinity]) | Single dose：pre-dose, at 2,5,8,12,25,45 minutes,1,2,4,8,12,24, 48,72,120 hours after-dose (When using Budesonide Powder for Inhalation, there is no need to monitor at 48, 72, and 120 hours after the end of administration)
  To characterize the pharmacokinetics of TQC3302 by assessment of area under the plasma concentration time curve from 0 extrapolated to infinity.
Time to reach maximum (peak) plasma concentration following drug administration (Tmax) | Single dose：pre-dose, at 2,5,8,12,25,45 minutes,1,2,4,8,12,24, 48,72,120 hours after-dose (When using Budesonide Powder for Inhalation, there is no need to monitor at 48, 72, and 120 hours after the end of administration)
  To characterize the pharmacokinetics of TQC3302 by assessment of time to reach maximum plasma concentration after single dosing.
Half-life (t1/2) | Single dose：pre-dose, at 2,5,8,12,25,45 minutes,1,2,4,8,12,24, 48,72,120 hours after-dose (When using Budesonide Powder for Inhalation, there is no need to monitor at 48, 72, and 120 hours after the end of administration)
  Terminal phase elimination half-life (T1/2) is the time required for half of the drug to be eliminated from the plasma.
Apparent volume of distribution (Vd/F) | Single dose：pre-dose, at 2,5,8,12,25,45 minutes,1,2,4,8,12,24, 48,72,120 hours after-dose (When using Budesonide Powder for Inhalation, there is no need to monitor at 48, 72, and 120 hours after the end of administration)
  Apparent volume of distribution of the TQC3302 in plasma.
Apparent clearance (CL/F) | Single dose：pre-dose, at 2,5,8,12,25,45 minutes,1,2,4,8,12,24, 48,72,120 hours after-dose (When using Budesonide Powder for Inhalation, there is no need to monitor at 48, 72, and 120 hours after the end of administration)
  Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the body.
Peak concentration (Cmax) after the first administration | Multiple dosing: at 2, 5, 8, 12, 25, 45 minutes, 1, 2, 4, 8, 12 hours after the first administration
  The Cmax is the maximum observed plasma concentration of study drug.
Time to reach maximum (peak) plasma concentration after the first administration (Tmax) | Multiple dosing: at 2, 5, 8, 12, 25, 45 minutes, 1, 2, 4, 8, 12 hours after the first administration
  To characterize the pharmacokinetics of TQC3302 by assessment of time to reach maximum plasma concentration after the first administration.
Half-life after the first administration | Multiple dosing: at 2, 5, 8, 12, 25, 45 minutes, 1, 2, 4, 8, 12 hours after the first administration
  Terminal phase elimination half-life (T1/2) is the time required for half of the drug to be eliminated from the plasma.
Area Under the Concentration-Time Curve From 0 to Last Observation after the first administration | Multiple dosing: at 2, 5, 8, 12, 25, 45 minutes, 1, 2, 4, 8, 12 hours after the first administration
  To characterize the pharmacokinetics of TQC3302 by assessment of area under the plasma concentration time curve from the first dose to a certain time point.
Area Under the Concentration-Time Curve From Zero to Infinity after the first administration | Multiple dosing: at 2, 5, 8, 12, 25, 45 minutes, 1, 2, 4, 8, 12 hours after the first administration
  To characterize the pharmacokinetics of TQC3302 by assessment of area under the plasma concentration time curve from 0 extrapolated to infinity
Peak concentration (Cmax) | Multiple dosing: at 2, 5, 8, 12, 25, 45 minutes, 1, 2, 4, 8, 12, 24 hours after the first dose, before Day 5, 6, 7, at 2, 5, 8,1 2, 25, 45 minutes, 1, 2 , 4, 8, 12, 24, 48, 72, 120 hours after Day 7 dose
  The Cmax is the maximum observed plasma concentration of study drug
Time to reach maximum (peak) plasma concentration following drug administration | Multiple dosing: at 2, 5, 8, 12, 25, 45 minutes, 1, 2, 4, 8, 12, 24 hours after the first dose, before Day 5, 6, 7, at 2, 5, 8,1 2, 25, 45 minutes, 1, 2 , 4, 8, 12, 24, 48, 72, 120 hours after Day 7 dose
  To characterize the pharmacokinetics of TQC3302 by assessment of time to reach maximum plasma concentration after multiple dosing
Area Under the Concentration-Time Curve From 0 to Last Observation (AUC [0-t]) | Multiple dosing: at 2, 5, 8, 12, 25, 45 minutes, 1, 2, 4, 8, 12, 24 hours after the first dose, before Day 5, 6, 7, at 2, 5, 8,1 2, 25, 45 minutes, 1, 2 , 4, 8, 12, 24, 48, 72, 120 hours after Day 7 dose
  To characterize the pharmacokinetics of TQC3302 by assessment of area under the plasma concentration time curve from the first dose to a certain time point
Area Under the Concentration-Time Curve From Zero to Infinity (AUC [0-infinity]) | Multiple dosing: at 2, 5, 8, 12, 25, 45 minutes, 1, 2, 4, 8, 12, 24 hours after the first dose, before Day 5, 6, 7, at 2, 5, 8,1 2, 25, 45 minutes, 1, 2 , 4, 8, 12, 24, 48, 72, 120 hours after Day 7 dose
  To characterize the pharmacokinetics of TQC3302 by assessment of area under the plasma concentration time curve from 0 extrapolated to infinity.
Area Under the Concentration-Time Profile From Time Zero to the Dosing Interval Tau | Multiple dosing: at 2, 5, 8, 12, 25, 45 minutes, 1, 2, 4, 8, 12, 24 hours after the first dose, before Day 5, 6, 7, at 2, 5, 8,1 2, 25, 45 minutes, 1, 2 , 4, 8, 12, 24, 48, 72, 120 hours after Day 7 dose
  Area Under the Concentration-Time Profile From Time Zero to the Dosing Interval Tau (AUCtau) of TQC3302 from the first dose to a certain time point.
Half-life (t1/2): Terminal phase elimination half-life (T1/2) is the time required for half of the drug to be eliminated from the plasma | Multiple dosing: at 2, 5, 8, 12, 25, 45 minutes, 1, 2, 4, 8, 12, 24 hours after the first dose, before Day 5, 6, 7, at 2, 5, 8,1 2, 25, 45 minutes, 1, 2 , 4, 8, 12, 24, 48, 72, 120 hours after Day 7 dose
  Terminal phase elimination half-life (T1/2) is the time required for half of the drug to be eliminated from the plasma.
Accumulation ratio based on peak concentration (Rac (Cmax)) | Multiple dosing: at 2, 5, 8, 12, 25, 45 minutes, 1, 2, 4, 8, 12, 24 hours after the first dose, before Day 5, 6, 7, at 2, 5, 8,1 2, 25, 45 minutes, 1, 2 , 4, 8, 12, 24, 48, 72, 120 hours after Day 7 dose
  Accumulation ratio based on peak concentration (Rac (Cmax))
Accumulation ratio based on AUC | Multiple dosing: at 2, 5, 8, 12, 25, 45 minutes, 1, 2, 4, 8, 12, 24 hours after the first dose, before Day 5, 6, 7, at 2, 5, 8,1 2, 25, 45 minutes, 1, 2 , 4, 8, 12, 24, 48, 72, 120 hours after Day 7 dose
  Accumulation ratio based on AUC

CONTACTS AND LOCATIONS:
Locations (1):
- China Japan Friendship Hospital Beijing, Beijing, Beijing Municipality, China